CLINICAL TRIAL: NCT01438736
Title: A Randomized Study to Evaluate the Predictive Impact of Using Cerazette Progestin Only Pill Before Nexplanon Insertion Regarding Bleeding Pattern
Brief Title: Is Cerazette Use Before Nexplanon Insertion Predictive for Bleeding Pattern?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VL-Medi Oy (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EudraCT 2011-001492-39; IIPS#39689 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Bleeding
Keywords: Focus:; preceding; desogestrel predicts; pattern of following; etonogestrel implant
MeSH Terms: conditions — Hemorrhage | interventions — Desogestrel; etonogestrel; Drug Implants

ARMS (2):
- Desogestrel, Etonogestrel (Experimental): Arm 1: 75 microgr desogestrel POP (cerazette) daily for 3 months followed by etonogestrel implant (Nexplanon, 68 mg etonogestrel) for following 6 months
  Interventions: Drug: Desogestrel 75 micrograms POP (Cerazette), Etonogestrel 68 mg implant (Nexplanon)
- Etonogestrel (Experimental): Arm 2: Women staring straight with Nexplanon implant for 6 months
  Interventions: Drug: Etonogestrel 68 mg subdermal implant

INTERVENTIONS:
Drug: Desogestrel 75 micrograms POP (Cerazette), Etonogestrel 68 mg implant (Nexplanon) — Desogestrel 75 micrograms POP daily for 3 monts, followed by etonogestrel 68 mg subdermal implant for following 6 months
  Arms: Desogestrel, Etonogestrel
Drug: Etonogestrel 68 mg subdermal implant — Etonogestrel 68 mg subdermal implant for 6 months
  Arms: Etonogestrel

SUMMARY:
The purpose of the study is to examine how well three months preceding use of Cerazette progestin only pill predicts the bleeding pattern during following Nexplanon implant use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, 18-40 years of age
* regular menstrual cycle (period 23-35 days)

Exclusion Criteria:

* -Immediate previous use of progestin only contraception within 2 months
* Known or suspected pregnancy
* Acute tromboembolic disorder
* Presence or history of hepatic disease, as long as the liver function values have not returned to normal
* Undiagnosed vaginal bleeding
* Known or suspected sex-steroid influenced malignancies (e.g. breast cancer)
* Hypersensitivity to the active substances or to any of the excipients of the medicines
* Pregnant or breast feeding within 6 weeks
* The use of other medicinal products that might interact with contraceptive steroids and affect the efficacy of contraceptives and/or might may lead to bleeding irregularities (especially medicines that induce the liver enzyme systems such as cytochrome P450). Examples of active substances are: phenytoin, phenobarbital, primidone, bosentan, carbamatzepine, rifampicin and medicinal products or herbal preparations containing ST.John's wort and to a lesser extend oxcarbazepine, topiramate, felbamate and griseofulvin.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
The total number of bleeding days per 90 days reference period in women using Cerazette before Nexplanon and in women starting Nexplanon without preceding POP | 9 months

SECONDARY OUTCOMES:
The number of bleeding episodes according to WHO definitions | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Dan Apter, Docent, Principal Investigator — VL-Medi Oy
Locations (1):
- VL Medi Oy, Helsinki, Finland